CLINICAL TRIAL: NCT02617108
Title: Randomized, Controlled Trial Comparing the Efficacy of Intrauterine Balloon and Postoperative Estrogen Therapy in the Prevention of Adhesion Reformation After Hysteroscopic Adhesiolysis
Brief Title: Intrauterine Balloon and Postoperative Estrogen Therapy in the Prevention of Adhesion Reformation After Hysteroscopic Adhesiolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Xiao Yu, Dr., Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FuXingH2
Record Dates: First submitted 2015-11-23; First posted 2015-11-30 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Uterine Septum
Keywords: uterine septum; intrauterine adhesions; Foley balloon
MeSH Terms: conditions — Septate Uterus; Gynatresia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foley balloon (Experimental): Foley balloon following TCRS: a Foley balloon with 4 ml of normal saline solution will be placed into the uterine cavity at the end of the operation for five days.
  Interventions: Device: Foley balloon
- control groups (No Intervention): control groups: women will not receive any therapy of the treatment (comparison group).
- postoperative estrogen therapy groups (Experimental): Subjects received postoperative hormone therapy as per the protocol in use in our center for Asherman Syndrome. Immediately after the operation, the subjects were started on a 3- month course of cyclical hormonal therapy, consisting of orally administrated oestradiol valerate 2-4mg/day for 21 days, orally administrated medroxyprogesterone acetate 8mg /day from day 12 to 21 of the oestradiol valerate therapy. The second treatment cycle started one week after the completion of the first cycle, and the third treatment cycle started one week after the second cycle.
  Interventions: Device: Foley balloon

INTERVENTIONS:
Device: Foley balloon — a Foley balloon with 4 ml of normal saline solution will be placed into the uterine cavity at the end of the operation for five days.
  Arms: Foley balloon; postoperative estrogen therapy groups

SUMMARY:
Patients who want to go TCRS will randomly divided 3 groups. In Group 1(100 patients), women received postoperative estrogen therapy. In Group 2 (100 patients), a Foley catheter with the balloon inflated with 4 ml of normal saline solution will be placed into the uterine cavity at the end of the operation for five days. In Group 3 (110 patients), women will not receive any of the treatment (comparison group). All subjects underwent two further hysteroscopy, one and three months after the initial surgery. At the second or third look hysteroscopy, the incidence of intra-uterine adhesion will be analyzed.

DETAILED DESCRIPTION:
The uterine septum (US) is the most common congenital uterine malformation, accounting for about 75% of Mullerian anomalies. Transcervical resection of septum (TCRS) has been shown in several cohort studies to improve outcome, although evidence from prospectively conducted randomized trial is lacking. TCRS is generally considered to be safe but there is a concern that it may be complicated by post-operative formation of intrauterine adhesions. Some investigators therefore recommend the use of postoperative adjuvant therapies with a view to preventing adhesion formation, as in the case of hysteroscopic surgery for Asherman syndrome. The adjuvant measures proposed include postoperative estrogen therapy, the placement of an intrauterine device (IUD) or Foley catheter in the uterine cavity. Unlike the case of Asherman syndrome in which these various adjuvant therapies are often used and appear to be of benefit, it is uncertain if any of these adjuvant measures are of benefit or necessary in the case TCRS. In this study, the investigators will compare the postoperative adhesion formation rates who will receive Foley catheter therapies 、postoperative estrogen therapy and those who will not receive any therapies to determine the usefulness of Foley catheter therapies in reducing postoperative adhesion formation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will go hysteroscopic transection of uterine septum between 2016 to 2017 at the Hysteroscopy Center, Fuxing Hospital;
* Patients willing to undergo followed hysteroscopy about 4 and 12 weeks after the surgery to assess the reformation of intrauterine adhesions;
* Written informed consent obtained.

Exclusion Criteria:

* ongoing pregnancy;
* Peroperative fever or infections;
* Malignancy;
* Precious pelvic inflammatory disease;
* Uterine fibroid (>3cm size);
* endometriosis;
* Contraindications for anesthesia;
* Not able to read and/or understand informed consent.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
A comparison of the presence and severity(American Fertility Society score) of intra-uterine adhesions at second look and third look hysteroscopy | 1 year
  the incidence and severity of adhesions (as measured according to the American Fertility Society scoring system) between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Tinchiu Li, Ph.D., Study Director — Chinese University of Hong Kong

REFERENCES:
- [Background] Hassan MA, Lavery SA, Trew GH. Congenital uterine anomalies and their impact on fertility. Womens Health (Lond). 2010 May;6(3):443-61. doi: 10.2217/whe.10.19. PMID 20426609
- [Background] Brucker SY, Rall K, Campo R, Oppelt P, Isaacson K. Treatment of congenital malformations. Semin Reprod Med. 2011 Mar;29(2):101-12. doi: 10.1055/s-0031-1272472. Epub 2011 Mar 24. PMID 21437824
- [Background] Lin X, Wei M, Li TC, Huang Q, Huang D, Zhou F, Zhang S. A comparison of intrauterine balloon, intrauterine contraceptive device and hyaluronic acid gel in the prevention of adhesion reformation following hysteroscopic surgery for Asherman syndrome: a cohort study. Eur J Obstet Gynecol Reprod Biol. 2013 Oct;170(2):512-6. doi: 10.1016/j.ejogrb.2013.07.018. Epub 2013 Aug 7. PMID 23932377
- [Background] Conforti A, Alviggi C, Mollo A, De Placido G, Magos A. The management of Asherman syndrome: a review of literature. Reprod Biol Endocrinol. 2013 Dec 27;11:118. doi: 10.1186/1477-7827-11-118. PMID 24373209